CLINICAL TRIAL: NCT05065775
Title: Intranasal Dexmedetomidine Pharmacokinetics on Patients Under General Anesthesia
Brief Title: Bioavailability of Intranasal Dexmedetomidine
Acronym: INDEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INDEX
Record Dates: First submitted 2021-10-01; First posted 2021-10-04 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Pharmacokinetics; Arthritis Knee; Arthritis of Hip; Anesthesia
Keywords: Intranasal; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexmedetomidine (Experimental): Single intranasal 100 µg bolus dose of dexmedetomidine
  Interventions: Device: Dexmedetomidine

INTERVENTIONS:
Device: Dexmedetomidine — Single intranasal dexmedetomidine dose of 100 µg. Intranasal dexmedetomidine will be administered shortly after induction of anesthesia using a mucosal atomization devise (LMA MAD Nasal™)
  Other Names: Dexdor

SUMMARY:
Aim of this study is to characterize the pharmacokinetics of dexmedetomidine in supine, anesthetized adult patients after intranasal dosing.

DETAILED DESCRIPTION:
To date, intranasal dexmedetomidine pharmacokinetics have not been studied before on anesthetized adult patients in supine position. As use of intranasal dexmedetomidine is growing, it is crucial to enhance knowledge of its pharmacokinetics.

Open, exploratory study design will be used. Study population will consist of patients coming to elective unilateral hip or knee arthroplasty under general anesthesia in Turku University Hospital, Salo unit. Thirty patients compatible with the inclusion and exclusion criteria will be entered into the study after receiving informed consent. Plasma concentrations of dexmedetomidine and other significant data will be collected prospectively.

Intranasal dexmedetomidine 100 ug will be administered shortly after induction of general anesthesia using a mucosal atomization (LMA MAD Nasal™) device, according to normal local protocol. Second cannula will be placed after patient is anesthetized, in order to obtain blood samples. Venous blood samples will be obtained immediately prior to administration of dexmedetomidine (baseline) and thereafter at 5, 15, 45 min and 1, 4 h into EDTA tubes for determination of dexmedetomidine, and possibly adrenaline and noradrenaline plasma concentrations.

Vital signs (heart rate, blood pressure and peripheral oxygen saturation) will be followed during the operation, as well as in the post anesthesia care unit according to the local protocol. Before patients will be admitted to the ward, they are expected to be appropriately arousable and have vital signs in normal limits.

ELIGIBILITY:
Inclusion Criteria:

* The patient is scheduled for elective unilateral total knee arthroplasty or hip arthroplasty under general anesthesia
* Fluent skills in finnish language (to understand the given information and to be able to give informed consent and communicate with the study personnel)
* Age between 35 and 80 years
* Weight between 50 and 100 kg
* ASA (American Society of Anesthesiologists) status 1-3
* Written informed consent from the patient

Exclusion Criteria:

* A previous history of intolerance to the study drug or related compounds and additives
* Disease or condition affecting patient's ability to give written informed consent
* Existing or recent significant disease possible affecting absorption, distribution, metabolism, excretion or response to the study drug
* History of cardiac disease (valvular insufficiency, severe left ventricular dysfunction) or abnormal ECG rhythm (bradycardia < 50/min, 2nd or 3rd degree atrio-ventricular block, pacemaker)
* Chronic opioid use or use of other analgesic adjuvants such as pregabalin, gabapentin, amitriptyline or duloxetine
* Participation in any other study concomitantly or within one month prior to the entry into this study
* Clinically significant abnormal findings in physical examination or laboratory screening
* Use of drugs or natural products known to cause enzyme induction or inhibition
* Pregnancy or breastfeeding
* Spinal anesthesia
* Preoperative systolic blood pressure <110 mmHg

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability (%) of intranasally given dexmedetomidine | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Panu Uusalo, MD, PhD, Principal Investigator — University of Turku and Turku University Hospital
Locations (1):
- Perioperative Services, Intensive Care and Pain Therapy, Turku University Hospital and University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No